CLINICAL TRIAL: NCT05657756
Title: Hand Dynamometer and Clinical Tests to Evaluate Neuromuscular Recovery in Atracurium vs Rocuronium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al Safwa University College (Other)
Responsible Party: Principal Investigator, Mohammed AbdulZahra Sasaa, principle investigator, Al Safwa University College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: hand dynamometer
Record Dates: First submitted 2022-11-04; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Neuromuscular Block Prolonged

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atracrium group (Other)
  Interventions: Device: Randomize clinical trial using hand dynamometer
- Rocoronium group (Other)
  Interventions: Device: Randomize clinical trial using hand dynamometer

INTERVENTIONS:
Device: Randomize clinical trial using hand dynamometer — Our research article involves 100 patients aged over 18 years old with ASAI&II divided into two groups, 50 patients will receive atracurium (0.5 mg/kg) and 30 patients receive Rocuronium (0.6 mg/kg). All of our patients will be undergoing elective laparoscopic surgery for cholecystectomy; the patients will randomly select to receive standard anesthesia induction with propofol (2 mg/kg), fentanyl (1-2 mcg/kg), and isoflurane 1.2 Mac, except muscle relaxant. Neuromuscular will monitoring by Train-of-Four (TOF) during surgery.

SUMMARY:
One of the common serious complications in the postoperative phase is Residual the neuromuscular blockade that confused the anesthesia medical team also patients may become uncomfortable, un ability to clear secretion, un-explanation of decreasing SPO2, increase respiratory effort and lead to an increase in the risk of respiratory complication. Most clinicians used clinical assessment to evaluate neuromuscular recovery such as a head lift for 5 seconds, Sustain leg lift, Tongue protrusion, teeth clenching, swallowing, Tidal volume 5 mL/kg, Handgrips Sustained for 5 seconds, and other clinical assessments in patients undergoing general anesthesia. A few studies have been discussing the utilization of hand dynamometers in the assessment of post-residual neuromuscular block. Our aim is to examine the neuromuscular recovery using a hand dynamometer after receiving Atracurium versus Rocuronium.

ELIGIBILITY:
Inclusion Criteria:

* all patient between 18-60 years old with ASAII under general anesthesia

Exclusion Criteria:

* all patient under 18 years old and over 60 years old
* prior administration of suxamethonium
* patient received magnesium, lithium, Quinidine, calcium channel blockers, local anesthesia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-10 (Estimated)

PRIMARY OUTCOMES:
100 patients were enrolled in our study, they are receiving muscle relaxants either Atracurium or rocuronium, and we recorded the muscle strength of the forearm in a postoperative location using an electronic hand dynamometer with a kilogram scale. | up to 6 months
  record the neuromuscular recovery using a hand dynamometer with a kilogram scale

CONTACTS AND LOCATIONS:
Locations (1):
- mohammed abdulzahra Sasaa, Najaf, Adala, Iraq

IPD SHARING:
Plan to Share IPD: No